CLINICAL TRIAL: NCT07264530
Title: The Relationship Between the Blockage of the Sacroiliac Joint (SI) and the Spasm of the Piriformis Muscle.
Brief Title: The Relationship of the Joint Blockage and Muscle Spasm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Malá Jitka, PhDr. Jitka Malá, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Svobodova, Piriformis
Record Dates: First submitted 2025-11-20; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: NO DECOMPENSATED ILLNESS; Muscle Cramps; Joint Dysfunction
Keywords: joint blockage; muscle spasm; muscle irritability
MeSH Terms: conditions — Muscle Cramp; Joint Diseases; Spasm

STUDY DESIGN:
Intervention Model Description: A group of suitable subjects (n=40) is divided into an experimental group and a control group (n=20). All subjects meet the study's inclusion criteria. All subjects undergo the same initial examination, including palpation of the piriformis muscle, joint play of the sacroiliac joint, and a visual analogue scale. The experimental group is treated with mobilisation techniques and left to rest for 30 minutes. The control group receives no mobilisation intervention and is only left to rest for 30 minutes. Subsequently, an exit examination identical to the entrance examination is performed. The results are entered into Excel tables and further processed using statistical methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental investigated group (Experimental): Group to which the mobilization technique will be applied to the sacroiliac joint according to "Cluster of Lasslet"
  Interventions: Procedure: Mobilization technique for sacroiliac joint
- Control non-investigated group (No Intervention): A control group that undergoes an initial examination but subsequently receives no therapy. After 30 minutes of quiet rest, it is examined again.

INTERVENTIONS:
Procedure: Mobilization technique for sacroiliac joint — The subject lies on their stomach, mobilization maneuvers are performed, a total of 4 maneuvers according to the recommended "Cluster of Lasslet" procedure for the sacroiliac joint.
  Arms: Experimental investigated group

SUMMARY:
An interventional study aimed at verifying the effect of sacroiliac joint blockage on changes in piriformis muscle tension. The study was conducted on 40 subjects, both male and female. Physical therapy methods were used to diagnose muscle tension as a diagnostic tool, along with a visual analogue scale. The intervention was performed using manual mobilisation techniques commonly used in clinical practice. The effectiveness was verified using the same physical therapy diagnostic tool as at the beginning. The entire research process is time-consuming, taking up to 1 hour per examinee.

DETAILED DESCRIPTION:
Objectives: The main aim of this study is to summarise current knowledge about the relationship between functional joint blockage and chained muscle spasm. To verify the relationship between sacroiliac joint blockage and piriformis muscle using combined therapy as a diagnostic tool, where the main parameter monitored will be the intensity of piriformis muscle irritability before and after sacroiliac joint mobilisation.

Methods: Measurements will be taken on a group of 40 subjects. The research sample consists of people aged 18-60, randomly divided into an experimental and a control group. All subjects underwent an initial palpation examination of the piriformis muscle, during which the level of pain was determined on a numerical pain scale. All subjects then underwent measurement of the piriformis muscle's irritability threshold using the "Beauty-line device 4000 Topline" device. The experimental group then underwent therapeutic intervention in the form of sacroiliac joint mobilisation using the "Cluster of Lasslet" technique. This was followed by 30 minutes of relaxation. The control group received no therapeutic intervention and only 30 minutes of relaxation between the initial and final examinations. Both groups then underwent the same final examination as at the beginning.

The investigators expect a change in piriformis muscle hypertonicity after sacroiliac joint mobilisation, including a reduction in pain in this muscle, at a statistical significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* palpation sensitivity of the piriformis muscle in the piriformis line,
* limited joint play of the sacroiliac joint,
* pain in the lower back, groin, perineum, buttocks, or hips, tenderness in the sacrum,
* pain or weakness during resisted abduction at 90° flexion in the hip joint,
* positive piriformis sign, positive Freiberg's test, positive Trendelenburg's test, or positive Pace's abduction test.
* At least 50% of the accompanying signs of sacroiliac joint blockage must be present in each subject.

Exclusion Criteria:

* acute (primarily infectious) diseases,
* persons in acute condition after an accident,
* persons recovering from an accident/illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-11-10 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Changing of piriformis muscle irritability | one hour at all
  After removing the sacroiliac joint blockage, the irritability threshold of the piriformis muscle increases and its painfulness decreases. The reduction in pain will be evident based on instrumental measurements using the Beauty-line device and palpation examination.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Petr, Doc., Study Chair — Charles University, Faculty of physical education and sport
Locations (1):
- Vokovice, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
not enough experience